CLINICAL TRIAL: NCT02094079
Title: Monitoring and Evaluation of the Levothyroxin Replacement Therapy in Pregnant Women
Brief Title: Monitoring and Evaluation of the Levothyroxin Replacement Therapy in Pregnant Women With Hypothyroidism
Status: Completed | Type: Observational
Sponsor: Birte Nygaard (Other)
Responsible Party: Sponsor-Investigator, Birte Nygaard, Birte Nygaard, md, phd, Herlev Hospital
Organization: Herlev Hospital (Other)
Other Study IDs: pregnant hypo
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Hypothyroidism
Keywords: hypothyroidism; pregnancy
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- L-T4 treated hypothyroid pregnant women: L-T4 treated pregnant women
  Interventions: Other: biomedical outcomes

INTERVENTIONS:
Other: biomedical outcomes — Evaluation of abnormal blodtests (evaluating thyroid function) from predefined control program

SUMMARY:
The aim of the study was to evaluate the clinical control program in patients with hypothyroidism during pregnancy (suggested in resent guidelines). Is it possible by monitoring the patients every 4. week during pregnancy to keep the thyroid function parameters within the recommended range?

A retrospective study of consecutive pregnant women with hypothyroidism followed at the outpatient clinic at the Endocrinology Unit, Herlev Hospital, Denmark during 2012. Patients selected through electronic medical system. Blood tests for the The hormone levels drawn from the laboratory of Clinical Biochemical Department, Herlev Hospital

ELIGIBILITY:
Inclusion Criteria:

* Consecutive pregnant women with L-T4 treated hypothyroidism followed at the outpatient clinic at the Endocrinology Unit, Herlev Hospital, Denmark during 2012

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A retrospective study of consecutive pregnant women with L-T4 treated hypothyroidism followed at the outpatient clinic at the Endocrinology Unit, Herlev Hospital, Denmark during 2012
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
number of patients with thyroid function parameters within the intended level | nine months

SECONDARY OUTCOMES:
number of complications during pregnancy | nine months

CONTACTS AND LOCATIONS:
Overall Officials: Birte Nygaard, MD, phd, Principal Investigator — Endocrine Unit O, Herlev Hospital, University of Copenahgen
Locations (1):
- Endocrine Unit O, Herlev Hospital, University of Copenhagen, Herlev, Denmark

REFERENCES:
- [Derived] Hubaveshka J, Michaelsson LF, Nygaard B. The dose of levothyroxine in pregnant women with hypothyroidism should be increased by 20-30% in the first trimester. Dan Med J. 2014 Dec;61(12):A4959. PMID 25441726